CLINICAL TRIAL: NCT02470806
Title: A Prospective, Randomized, Comparative Effectiveness Study of a Single-Use, Negative Pressure Wound Therapy System (PICO) Versus a Traditional Negative Pressure Wound Therapy System (tNPWT) in the Treatment of Lower Extremity Ulcers
Brief Title: Single-Use Negative Pressure Wound Therapy System vs. Traditional Negative Pressure Wound Therapy System (tNPWT)
Acronym: NPWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CE-052PIC
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Venous Leg Ulcers; Diabetic Foot Ulcers
Keywords: Venous leg ulcer; ulcer; venous stasis; compression; diabetic foot ulcers; dfu; vlu
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICO System (Experimental): Negative Pressure Wound Therapy (NPWT) at 80mmHg (nominal) +/- 20 mmHg to the wound surface
  Interventions: Device: PICO System
- tNPWT System (Active Comparator): Traditional NPWT (tNPWT) from -25 mmHg and up to -200 mmHg; intensity settings of either low, medium and high; delivery modes of continuous or intermittent. The pressure, intensity and delivery settings will be left to the Investigator's discretion at each study treatment visit.
  Interventions: Device: tNPWT System

INTERVENTIONS:
Device: PICO System — Negative Pressure Wound Therapy (NPWT) at 80mmHg (nominal) +/- 20 mmHg to the wound surface
  Arms: PICO System
Device: tNPWT System — NPWT from -25 mmHg and up to -200 mmHg; intensity settings of either low, medium and high; delivery modes of continuous or intermittent. The pressure, intensity and delivery settings will be left to the Investigator's discretion at each study treatment visit.
  Arms: tNPWT System

SUMMARY:
The aim of this study is to compare the clinical efficacy of two types of NPWT systems; the traditional negative pressure wound therapy (tNPWT) system and the single-use negative pressure wound therapy (PICO) system.

DETAILED DESCRIPTION:
The two types of NPWT systems include the tNPWT system that has successfully completed a coding verification request with CMS and has the following capabilities (e.g., range of negative pressure, connective tubing, canister, foam or gauze filler, and approved for home use), and a portable, canister-less, battery operated, disposable PICO system to see if there are any observed differences with regard to the clinical efficacy of the two devices.

ELIGIBILITY:
INCLUSION CRITERIA:

* Provide informed consent
* Age ≥ 18 years and of either sex
* Willing to comply with protocol instructions, including allowing all study assessments
* Have a Venous Leg Ulcer (VLU) between the knee and ankle (at or above the malleolus), with a surface area ≥ 2.0 cm2 and ≤ 36.0 cm2
* Target ulcer duration ≥ 4 weeks but ≤ 104 weeks (24 months)
* Have a Diabetic Foot Ulcer (DFU) present on any part of the plantar or dorsum surface of the foot, with a surface area ≥ 0.5 cm2 and ≤ 10.0 cm2
* Target ulcer involves a full thickness skin loss, but WITHOUT exposure of tendon, muscle, or bone
* Target ulcer duration ≥ 4 weeks but ≤ 52 weeks (12 months)
* Acceptable state of health and nutrition

EXCLUSION CRITERIA

* Therapy with another investigational agent within thirty (30) days of Screening, or during the study Ulcers which are deemed as highly exuding, per the Investigator's discretion.
* Current diagnosis of osteomyelitis at the target wound location that is not currently receiving treatment [Documented history of resolved osteomyelitis is allowed].
* Subjects with a VLU: Refusal of or inability to tolerate compression therapy.
* Clinical evidence of target ulcer infection
* Current systemic therapy with cytotoxic drugs.
* Current therapy with chronic (> 10 days) oral corticosteroids.
* Previous treatment with NPWT device or hyperbaric oxygen within 7 days of screening.
* Malignancy in the target ulcer, or history of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Weymann, MD, MBA, Study Chair — Smith & Nephew, Inc.
Locations (17):
- United States (15):
  - ILD Consulting, Inc., Carlsbad, California
  - Valley Foot & Ankle Specialty Providers, Fresno, California
  - The Sun Healthcare & Surgery Group, Martinez, California
  - Center for Clincial Research, San Francisco, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - University of Miami, Miami, Florida
  - NW University Feinberg School of Medicine, Chicago, Illinois
  - Rosalind Franklin University of Med & Science, North Chicago, Illinois
  - Ochsner Health System, New Orleans, Louisiana
  - Rubin Institute for Advanced Orthopedics, Baltimore, Maryland
  - Advanced Foot & Ankle, Las Vegas, Nevada
  - Center for Advanced Wound Care, Wyomissing, Pennsylvania
  - Acclaim Bone & Joint, Fort Worth, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Carilion Clinic, Roanoke, Virginia
- Canada (2):
  - The Mayer Institute, Hamilton, Ontario
  - Centre podiatrique et soins des plaies, Boucherville, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- PICO System: Subjects randomized to receive the PICO system applied to the target ulcer area over the 12-week treatment period from Baseline.
- tNPWT System: Subjects randomized to receive the tNPWT system applied to the target ulcer area over the 12-week treatment period from Baseline.
Period: Overall Study
Arm/Group | PICO System | tNPWT System
Started | 80 | 84 (The Safety analysis included 164, ITT was 161, and Per Protocol was 115 subjects (total both arms).)
Completed | 62 | 42
Not Completed | 18 | 42
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 5 | 2
Not completed — Protocol Violation | 4 | 11
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 3 | 10
Not completed — Lack of Efficacy | 5 | 15

BASELINE CHARACTERISTICS:
Population: The Safety analysis included all enrolled subjects (N=164), however, 3 subjects did not complete a follow-up visit and thus were excluded from all Baseline and Outcome Measure analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | PICO System | tNPWT System | Total
Number analyzed (Participants) | 80 | 81 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (14.7) | 60.4 (11.9) | 61.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 48 | 54 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 77 | 79 | 156
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 12 | 20
  White | 67 | 67 | 134
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 5 | 7
  United States | 78 | 76 | 154
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 33.7 (8.8) | 33.9 (9.0) | 33.8 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Ulcer Area From Baseline to the End of the Treatment Period
Description: Ulcer area was photographed in order to determine the measurements of the post-debridement ulcer area (cm^2 and total percentage [%]) using the ARANZ Silhouette wound imaging and measurement device.
Time Frame: Baseline through 12 weeks
Population: The Per-Protocol (PP) population was used to analyze outcome measure data and included all subjects who were randomized, met inclusion/exclusion criteria, had not discontinued treatment within the first 9 weeks (-1 day), and had no significant protocol deviations.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | PICO System | tNPWT System
Number analyzed (Participants) | 64 | 51
cm^2
  Baseline wound area | 6.2 (5.9) | 7.8 (6.3)
  Final wound area | 0.7 (1.8) | 3.8 (6.7)
  Change in wound area | -5.5 (5.4) | -4.0 (6.2)
Statistical Analysis 1: Comparison: PICO System vs tNPWT System; Percentage change in wound area from Baseline to end of 12-week treatment period (PP population - all wounds); Test type: Non-Inferiority — Stepwise regression method - Primary efficacy analysis, difference between treatment groups in percentage change in wound area from baseline visit to end of 12-week treatment period for the PP population; p = 0.001, Stepwise regression

2. Primary Outcome: Percentage Change in Ulcer Area From Baseline to the End of the Treatment Period
Description: Ulcer area was photographed in order to determine the measurements of the postdebridement ulcer area (cm^2 and total percentage [%]) using the ARANZ Silhouette wound imaging and measurement device.
Time Frame: Baseline through 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change in wound area
Arm/Group | PICO System | tNPWT System
Number analyzed (Participants) | 64 | 51
Percentage of change in wound area | -88.7 (24.1) | -58.6 (63.5)

3. Secondary Outcome: Change in Target Ulcer Depth Following Treatment With Either PICO or tNPWT From Baseline Over the 12-week Treatment Period
Description: Ulcer area was analyzed for depth measurement in millimeters (mm), volume measurement in cubic centimeters (cm^3), and percentage change (%) including terms for treatment, baseline depth, baseline volume, wound type, pooled sites, and wound duration using the ARANZ Silhouette wound imaging and measurement device.
Time Frame: Baseline through 12 weeks
Population: Change in wound depth over 12-week treatment period by treatment group (PP population - all wounds)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PICO System | tNPWT System
Number analyzed (Participants) | 64 | 51
mm
  Baseline wound depth | 4.0 (6.8) | 2.4 (1.3)
  Final wound depth | 0.6 (1.1) | 1.5 (2.1)
  Change in wound depth | -3.4 (7.1) | -0.9 (1.9)

4. Secondary Outcome: Change in Target Ulcer Volume Following Treatment With Either PICO or tNPWT From Baseline Over the 12-week Treatment Period
Description: as for outcome 3
Time Frame: Baseline through 12 weeks
Population: Change in wound volume over 12-week treatment period by treatment group (PP population - all wounds)
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | PICO System | tNPWT System
Number analyzed (Participants) | 64 | 51
cm^3
  Baseline wound volume | 0.3 (0.3) | 0.3 (0.3)
  Final wound volume | 0.2 (0.5) | 0.1 (0.3)
  Change in wound volume | -0.3 (0.3) | 0 (0.4)

5. Secondary Outcome: Percentage Change in Target Ulcer Depth and Volume Following Treatment With Either PICO or tNPWT From Baseline Over the 12-week Treatment Period
Description: as for outcome 3
Time Frame: Baseline through 12 weeks
Population: Percentage change in wound depth and volume over 12-week treatment period by treatment group (PP population - all wounds)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PICO System | tNPWT System
Number analyzed (Participants) | 64 | 51
percent change
  Percentage change from baseline in wound depth | -68.8 (59.4) | -38.8 (71.3)
  Percentage change from baseline in wound volume | -98.0 (8.1) | -10.1 (207.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline through 12 weeks of treatment or study withdrawal, whichever came first.
Arm/Group | PICO System | tNPWT System
All-Cause Mortality (participants affected / at risk) | 2/80 | 0/84
Serious Adverse Events (participants affected / at risk) | 6/80 | 8/84
Other Adverse Events (participants affected / at risk) | 65/80 | 57/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PICO System (N=80) | tNPWT System (N=84)
Abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 (0) | 2 (2)
Diastolic heart failure (Cardiac disorders) | 0 (0) | 2 (2) — Acute-on-chronic
Fluid collection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Thigh
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psychiatric evaluation (Psychiatric disorders) | 1 (1) | 0 (0)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Ulcer increased in size (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PICO System (N=80) | tNPWT System (N=84)
Target ulcer increase in size > 75% from Baseline (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Excessive maceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — The AE was considered mild.
Excessive intermittent maceration right plantar forefoot target ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Intermittent events caused intermittent stoppages in therapy. The AE was considered mild.
Deep venous thrombosis right lower leg (Vascular disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Right lateral midfoot blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Increased peri-wound maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Target venous leg ulcer maceration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) — The AE was considered mild.
Subject could not tolerated NPWT, it was uncomfortable for the subject (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Peri-ulcer tissue very macerated (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — The AE was considered moderate.
Left foot target ulcer cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Methicillin-resistant Staphylococcus aureus infection (Infections and infestations) | 1 (1) | 0 (0) — The AE was considered mild.
Target ulcer infection (Infections and infestations) | 2 (2) | 3 (3) — The AE was considered moderate.
Cellulitis to left 3rd interspace (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Subjective complaint of ulcer pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Abrasion at 10 o'clock from left distal dorsal TMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — The AE was considered mild.
Cellulitis of left plantar medial midfoot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Urinary tract infection (Renal and urinary disorders) | 1 (2) | 1 (1) — The AE was considered mild.
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Right ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Right thigh fluid collection with right groin incision site related drainage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Venous stasis ulcer pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
High blood pressure (Vascular disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Allergic contact dermatitis of the right leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Left ankle swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Left sole wound infection (Infections and infestations) | 1 (1) | 0 (0) — The AE was considered moderate.
Allergic contact dermatitis of skin surrounding right foot ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) — The AE was considered moderate.
Stasis dermatitis, xerosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — The AE was considered mild.
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Erythema intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Peri-wound maceration on left foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Peri-wound margin increase in maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Wound increased in size (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Regression in wound - size of wound increased by more than 75% from last visit (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Peri-wound maceration on right foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — The AE was considered mild.
Wound macerated (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Pressure-related pain from negative pressure (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Peri-wound maceration (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (12) — The AE was considered mild.
Pruritus RLE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Blistered skin right lower extremity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Probable osteomyelitis right foot at target ulcer (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Excoriations, maceration peri-wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Macerated skin left leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Redness, swelling, and discomfort right leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Progressive disease - worsening of target ulcer causing subject to be discontinued from study (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Worsening of coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Fall (General disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Infected pimple on face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
DFU (target ulcer) progressive disease (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Target wound pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
New non-target ulcer near target ulcer on right shin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
New non-target ulcer near target ulcer 0.5 cm in size (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Target wound pain decreased (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Debridement pain on target ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Right upper quadrant/back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Non-target ulcer on lateral side of left leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Multiple skin tears around target ulcer site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Water blister on medial side of left leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Skin tear adjacent to target ulcer on left leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Three skin tears 2 cm away from target wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Non-target wound on right lateral ankle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Maceration (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (7) — The AE was considered mild.
Two skin tears away from target wound (anterior) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Two skin tears posterior to left leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Multple skin tears from target wound anterior left leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Non-target wound on left leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Small irritations around where dressing puts pressure on left leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Left medial ankle venous leg ulcer bacterial colonization of wound bed (Infections and infestations) | 0 (0) | 1 (1) — The AE was considered mild.
Peri-wound skin irritated (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Right target ulcer larger (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Venous ulcer right leg malleolus increase in wound size (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Cellulitis of right foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Wet gangrene 4th digit left foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Peri-wound inflammation target leg left VLU (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Large amount of drainage from target ulcer, left leg calf (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Foot edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Foot blistering on dorsal and medial surface (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Suspected non-target ulcer infection (Infections and infestations) | 1 (1) | 0 (0) — The AE was considered moderate.
Formed a blister on anterior shin from tNPWT bridge (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Venous leg ulcer on left lateral leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Ulcer on dorsal portion of right foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Worsening of left ankle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Abdominal pain, epigastric (Gastrointestinal disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Episode of recurrent major depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Osteomyelitis of ankle/foot (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — The AE was considered moderate.
Bilateral lower extremity edema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — The AE was considered mild.
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — The AE was considered mild.
Acute urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Complication of Foley catheter (Renal and urinary disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Acute abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Edema, unspecified (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Suspected cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Intermittent burning/stabbing pain x1 week (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) — The AE was considered mild.
Left side of nose epidermal inclusion cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Left lower abdomen epidermal cyst inflamed (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Left lower leg swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Prolonged pain at target ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) — The AE was considered mild.
Bone exposure at target ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Wound undermining < 2 cm (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — The AE was considered mild.
Bulla right foot lateral side (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Progressive disease - wound size met the definition of progressive disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Burning pain in foot of target ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Target ulcer pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Scrotal edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — The AE was considered mild.
Contact dermatitis on left foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — The AE was considered mild.
Acute on chronic congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Wound infection (Infections and infestations) | 1 (1) | 0 (0) — The AE was considered mild.
Bone necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Left ankle and lower leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Body rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Additional ulcer left ankle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Right mid thigh lacerations (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Increased maceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Fracture of vertebral disk (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The AE was considered moderate.
Reopening of ulcers on target limb (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Worsening of recurring non-target ulcers on target limb (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered moderate.
Worsening of target ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Redness, skin breakdown to target limb (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — The AE was considered mild.
Swelling of the right foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The AE was considered mild.

LIMITATIONS AND CAVEATS:
There were no known limitations or caveats reported during this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT02470806/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT02470806/SAP_001.pdf